CLINICAL TRIAL: NCT05965635
Title: The Uninfected Ixodes Scapularis Human Tick Challenge Model
Acronym: TICK ME
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other)
Responsible Party: Principal Investigator, prof. J.W.R. Hovius, MD, PhD, PI, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: NL81259.018.22
Record Dates: First submitted 2023-03-28; First posted 2023-07-28 (Actual); Last update posted 2023-07-28 (Actual); Status verified 2023-03

CONDITIONS: Tick Bites; Tick Immunity
Keywords: Tick bites; Ixodus scapularis; Tick Challenge model; Tick borne diseases; Tick immunity
MeSH Terms: conditions — Tick Bites; Tick-Borne Diseases

STUDY DESIGN:
Intervention Model Description: Single centre, experimental study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental (Experimental)
  Interventions: Other: Ixodus scapularis nymphs

INTERVENTIONS:
Other: Ixodus scapularis nymphs — Tick challenge

SUMMARY:
An innovative way to prevent multiple tick-borne diseases is an anti-tick vaccine, i.e. targeting the vector to prevent transmission of pathogens from the tick to the host. The rationale for an anti-tick vaccine stems from a phenomenon coined tick immunity. This study aims to show proof of concept that humans indeed develop immunity to ticks. Therefore subjects will be challenged three to four times with ticks reared in colony from a designated laboratory and that are exhaustively tested negative for various known tick-borne pathogens. Several tick feeding parameters will be evaluated to assess the development of tick immunity in the subjects. To this end, a total amount of ten ticks per challenge will be placed under a dressing placed on the forearm. The primary study endpoint is the tick feeding phenotype. Secondary parameters are signs of an immune response in the host; itch, redness, or other signs of a (local) immune response (blood and skin biopsies). All parameters, except for the skin biopsies, will be collected/evaluated after each tick challenge.

DETAILED DESCRIPTION:
This will be an, single centre, experimental study. The design of the study is similar to a human challenge trial, with the important exception that the subjects in this study are not experimentally infected with a pathogen, but are exposed to well-characterized laboratory-reared uninfected nymphal Ixodes scapularis ticks.

Seven healthy human volunteers of >18 years old who have no history of known tick-bites or tick-borne diseases will be recruited. Subjects will undergo three to four tick challenges, consisting of five to six days per challenge with two weeks between the consecutive challenges. The total duration of participation is approximately five months for each subject. By making use of ticks from a laboratory-reared tick colony that have been, and are being, used in xenodiagnosis and tick challenge models in the USA and that are well tolerated minimizing the risks of the tick challenges. Regardless, the tick challenge can cause some discomfort because of possible local reactions and because the dressing must be kept dry for five to six days. The risk of infection with a tick-borne pathogen is negligible due to the fact that these ticks are exhaustively tested for various known tick-borne pathogens. Finally, risks are considerated of development of a red meat allergy or other allergic reactions negligible because no clear associations are known of I. scapularis ticks and red meat allergy. No serious adverse events (such as human infections or red meat allergy) have resulted from more than >100 challenges in the United States using this tick colony. There are no direct benefits of participation.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18 years and older;
* Negative Borrelia VlsE1/pepC10 ELISA.

Exclusion Criteria:

* Known history of tick bites;
* Positive Borrelia serology (VlsE1/PepC10 ELISA);
* Known history or current suspicion on any tick-borne disease;
* Chronic skin condition affecting the arm skin;
* Inability to maintain the dressing for any reason;
* Known immunodeficiency or autoimmune disease;
* Use of systemic immunomodulating drugs or chemotherapy, current or in the past;
* Chronic use of antibiotics;
* Unable to give informed consent or do not have a thorough command of the Dutch language;
* Refusal to participate in specimen collection and storage for future study related use;
* Pregnant or breastfeeding women;
* Not willing to use adequate contraception during the study period;
* Red meat allergy (both medically confirmed and self-reported);
* Use of investigational therapy and devices during the time of the study;
* Any other condition that, in the opinion of the investigator, would make the patient unsuitable for enrolment or could interfere with the patient participating in and completing the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 7 (Estimated)
Dates: Start 2023-07 (Estimated); Primary Completion 2024-07 (Estimated); Study Completion 2024-07 (Estimated)

PRIMARY OUTCOMES:
Tick weight | Up to 1 week
  Tick weight in mg
Tick feeding molting success | Up to 1 week
  Molting success rate
Tick survival | Up to 1 week
  tick survival rate
Tick attachment | Up to 1 week
  tick attachment rate

SECONDARY OUTCOMES:
Signs of an immune response in the host: Itch | Up to 1 week
  Itch
Signs of an immune response in the host: redness | Up to 1 week
  Redness
Signs of an immune response in the host: other | 3 weeks
  Other signs of a local immune response (in blood)
Signs of an immune response in the host: biopsies | 9 weeks
  Other signs of a local immune response (in skin biopsies)

CONTACTS AND LOCATIONS:
Locations (1):
- AUMC location AMC, Amsterdam-Zuidoost, North Holland, Netherlands

IPD SHARING:
Plan to Share IPD: No